CLINICAL TRIAL: NCT04618770
Title: A Prospective, Post-market, Multi-center Evaluation of the Clinical Outcomes of the Triathlon Total Knee System Using the Triathlon PSR Tibial Insert
Brief Title: Triathlon PSR Outcomes Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Sponsor decision due to lack of enrolment
Sponsor: Stryker Orthopaedics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 103
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Results first posted 2023-11-07 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Arthroplasty; Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Triathlon PSR Tibial Insert (Other): Cases receiving a Triathlon Total Knee with the Triathlon PSR Tibial Insert
  Interventions: Device: Triathlon PSR Tibial Insert

INTERVENTIONS:
Device: Triathlon PSR Tibial Insert — The Triathlon PSR Tibial Insert is intended to be used as a component in primary TKA and is designed to reduce rotational constraint at deep flexion.

SUMMARY:
This study is a prospective, open-label, post-market, non-randomized, multi-center clinical evaluation of the Triathlon Total Knee System using the Triathlon PSR Tibial Insert for primary total knee arthroplasty (TKA) in a consecutive series of patients who meet the eligibility criteria. The SF-36 score of subjects receiving the Triathlon Total Knee with the Triathlon PSR insert is expected to be comparable with that of subjects receiving historical Triathlon PS cemented constructs.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has signed an IRB/EC approved; study specific Informed Patient Consent Form.
2. Patient is a male or non-pregnant female, skeletally mature, age 18-75 years at time of study device implantation.
3. Patient has a diagnosis of Non-Inflammatory Degenerative Joint Disease (NIDJD).
4. Patient is a candidate for primary cemented total knee replacement.
5. Patient is willing and able to comply with postoperative scheduled clinical and radiographic evaluations and rehabilitation.

Exclusion Criteria:

1. Patient has a Body Mass Index (BMI) > 45.
2. Patient is already participating in the study for a contralateral total knee replacement.
3. Patient has a diagnosis of avascular necrosis or inflammatory arthritis.
4. Patient has an active or suspected latent infection in or about the affected knee joint at time of study device implantation.
5. Patient has any mental or neuromuscular disorder which would create an unacceptable risk of prosthesis instability, prosthesis fixation failure, or complications in postoperative care.
6. Patient has a compromised bone stock which cannot provide adequate support to the prosthesis.
7. Patient is immunologically suppressed or receiving steroids in excess of normal physiological requirements (e.g. > 30 days).
8. Patient is diagnosed with lumbar radicular pain.
9. Patient has severe instability of the knee joint secondary to the absence of collateral ligament integrity and function.
10. Patient has a known sensitivity to device materials.
11. Patient is a prisoner.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2021-02-08 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- OrthoCarolina, Charlotte, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Triathlon PSR Tibial Insert
Started | 37
Completed | 0
Not Completed | 37
Not completed — Censored from Analysis | 12
Not completed — Early Termination | 25

BASELINE CHARACTERISTICS:
Population: Participants
Arm/Group | Triathlon PSR Tibial Insert
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.96 (6.22)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9
  Male | 16
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Mean SF-36 Physical Component Score
Description: The SF-36 is a 36-item patient completed questionnaire to measure general health and well-being. It includes physical and mental status component sub scores; each ranging from 0-100. Low values represent a poor health state and high values represent a good health state.
Time Frame: pre-operative, 6 weeks, 1 year
Population: Subjects data collection through 1 year as study was early terminated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Triathlon PSR Tibial Insert
Number analyzed (Participants) | 25
score on a scale
  Physical SF-36-Preop | 34.17 (8.45)
  Physical SF-36-6 weeks: number analyzed (Participants) | 24
  Physical SF-36-6 weeks | 34.10 (9.10)
  Physical SF-36-1 year: number analyzed (Participants) | 6
  Physical SF-36-1 year | 41.85 (10.14)
  Mental SF-36-Preop | 55.87 (9.72)
  Mental SF-36-6 weeks: number analyzed (Participants) | 24
  Mental SF-36-6 weeks | 54.40 (9.07)
  Mental SF-36-1 year: number analyzed (Participants) | 6
  Mental SF-36-1 year | 53.44 (9.59)

2. Secondary Outcome: EuroQol-5 Dimension (EQ-5D)
Description: The EuroQol-5 Dimension (EQ-5D) is a subject-completed questionnaire designed to assess subject health state values. The EQ-5D consists of 2 areas; EQ-5D descriptive system and the visual analogue scale (VAS). The EQ-5D descriptive system comprises the following five dimensions: mobility self care, usual activities, pain/comfort and anxiety/depression. Each dimension has 3 levels indicating no problems, some problems or extreme problems. The index values on a scale between -1 (low) and 1 (high) are showing the average health status according to the 5 dimensions: A low score shows worse health and a high score shows better health.
  With the EQ VAS the respondents can report their perceived health status with a grade ranging from 0 (the worst possible health status) to 100 (the best possible health status).
Time Frame: PreOp, 6 week, 1 year
Population: Subjects data collection through 1 year as study was early terminated.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Triathlon PSR Tibial Insert
Number analyzed (Participants) | 25
score on a scale
  Descriptive EQ-5D-PreOp | 0.71 (0.14)
  Descriptive EQ-5D-6 weeks: number analyzed (Participants) | 24
  Descriptive EQ-5D-6 weeks | 0.76 (0.11)
  Descriptive EQ-5D-1 year: number analyzed (Participants) | 6
  Descriptive EQ-5D-1 year | 0.80 (0.13)
  VAS EQ-5D-PreOp | 80.00 (14.35)
  VAS EQ-5D-6 weeks: number analyzed (Participants) | 24
  VAS EQ-5D-6 weeks | 81.50 (12.50)
  VAS EQ-5D-1 year: number analyzed (Participants) | 6
  VAS EQ-5D-1 year | 88.33 (9.56)

3. Secondary Outcome: Range of Motion
Description: Range of Motion evaluates how much the knee can be bent and straightened. The normal range of motion is typically 0 to 135 degrees.
Time Frame: PreOp, 6 weeks, 1 year
Population: Subjects data collection through 1 year as study was early terminated.
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Triathlon PSR Tibial Insert
Number analyzed (Participants) | 25
degrees
  ROM-PreOp | 116.32 (7.92)
  ROM-6 weeks: number analyzed (Participants) | 24
  ROM-6 weeks | 111.08 (10.70)
  ROM-1 year: number analyzed (Participants) | 5
  ROM-1 year | 122.00 (5.70)

4. Secondary Outcome: Survivorship of Triathlon PSR Insert
Description: All-cause survivorship of the Triathlon PSR Tibial Insert will be evaluated through 10 year.
Time Frame: 1 Year
Population: At timepoint of termination, all enrolled and active subjects had the study device implanted.
Measure: Count of Participants; unit: Participants
Arm/Group | Triathlon PSR Tibial Insert
Number analyzed (Participants) | 25
Participants | 25

ADVERSE EVENTS:
Time Frame: 1 year
Description: No difference of adverse event definition.
Arm/Group | Triathlon PSR Tibial Insert
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of subjects analyzed due to lack of enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-04-13): https://cdn.clinicaltrials.gov/large-docs/70/NCT04618770/Prot_SAP_000.pdf
  • Informed Consent Form (2021-04-13): https://cdn.clinicaltrials.gov/large-docs/70/NCT04618770/ICF_002.pdf